CLINICAL TRIAL: NCT02179125
Title: Identifying REsponders and Exploring Mechanisms of ACTION of the Endobronchial Coil Treatment for Emphysema
Acronym: REACTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Dirk-Jan Slebos, MD PhD, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REACTION; NL49716.042.14 (Other: ABR-Form)
Record Dates: First submitted 2014-06-25; First posted 2014-07-01 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Endobronchial treatment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bronchoscopic LVR-coil treatment (Experimental): Bronchoscopic lung volume reduction with coil treatment
  Interventions: Device: RePneu Lung Volume Reduction Coil System

INTERVENTIONS:
Device: RePneu Lung Volume Reduction Coil System — Bronchoscopic lung volume reduction treatment with Coils.

SUMMARY:
Rationale: The PneumRx RePneu Lung Volume Reduction Coil (RePneu LVR-coil) is a bronchoscopic lung volume reduction treatment designed to compress the areas of lung parenchyma most damaged by emphysema. The LVRC treatment was found to be feasible, safe and effective in previous studies. However, patient-based outcomes besides quality of life questionnaires are hardly measured after intervention treatments for COPD. Furthermore, the exact underlying physiological mechanism of the LVR-coil treatment is unknown. Another aspect of the treatment which we to date do not fully understand is which group of patients benefit of the treatment and which group of patients do not, this knowing that the responder rate is already about 60%.

Objective: The objectives of the study are to gain more knowledge on 1) the effect of the LVRC treatment on patient-based outcomes like physical activity, 2) the underlying physiological mechanism of the treatment, 3) the predictors of response to the treatment at baseline, and 4) on a targetted treatment number of coils to be placed per lung using lung compliance.

Study design: This study is a non-randomised open label multi-center intervention study.

Study population: The study population exists of adult patients with severe emphysema with no other treatment options left besides surgical procedures.

Intervention: Bilateral bronchoscopic lung volume reduction treatment with RePneu coils.

Main study parameters/endpoints: The main study endpoint is the change in physical activity between baseline and 3 months follow-up after the second treatment. The secondary endpoints are the changes between baseline and 3 months follow-up after the second treatment in: patient reported outcomes of the treatment, dynamic lung hyperinflation, static lung volumes, lung compliance, diaphragm function, lung perfusion, systemic inflammation and small airways function.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The LVR Coil has been designed to be as safe as possible. It was shown that the risks associated with the LVRC system are largely attributable to the bronchoscopic procedure itself rather than to the device per se. Therefore, it appears that the LVRC device itself does not appreciably increase the risk of serious adverse events beyond the risk of undergoing a bronchoscopy procedure or simply having emphysema. Currently, this treatment is not commercially available in the Netherlands and study participants will have to visit the hospital multiple times. Previous studies have shown that the treatment has beneficial effect for the patient, however not all patients respond. Part of this new study is to try to identify which group of patients respond to the treatment and which patients do not. Therefore, it is possible that a patient will not receive any benefits from the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of COPD
2. FEV1%pred <45% and FEV1/FVC <60%
3. RV/TLC >55%
4. TLC%pred >100% AND RV%pred >175%
5. Dyspnea scoring ≥2 on mMRC scale of 0-4.
6. Stopped smoking for at least 6 months prior to entering the study.
7. Completed a pulmonary rehabilitation program within 6 months prior to treatment and/or regularly performing maintenance respiratory rehabilitation if initial supervised therapy occurred more than 6 months prior to baseline testing.
8. Received Influenza vaccinations consistent with local recommendations and/or policy.
9. Read, understood and signed the Informed Consent form.

Exclusion Criteria:

1. Subject has co-morbidities that may significantly reduce subject's ability to improve exercise capacity (e.g., severe arthritis, planned knee surgery) or baseline limitation on 6MWT is not due to dyspnea.
2. Subject has severe gas exchange abnormalities as defined by: PaCO2 >8.0 kPa and/or PaO2 < 6.0 kPa (on room air).
3. Subject has a history of recurrent clinically significant respiratory infections, defined as 3 or more hospitalizations for respiratory infection during the year prior to enrolment.
4. Subject has severe pulmonary hypertension defined by right ventricular systolic pressure >45 mm Hg via echocardiogram.
5. Subject has an inability to walk >140 meters in 6 minutes.
6. Subject has evidence of other severe disease (such as, but not limited to, lung cancer or renal failure), which in the judgment of the investigator may compromise survival of the subject for the duration of the study.
7. Subject is pregnant or lactating, or plans to become pregnant within the study timeframe.
8. Subject has an inability to tolerate bronchoscopy under conscious sedation or general anaesthesia.
9. Subject has clinically significant bronchiectasis.
10. Subject has giant bullae >1/3 lung volume.
11. Subject has had previous LVR surgery, lung transplantation or lobectomy.
12. Subject has been involved in pulmonary drug or device studies within 30 days prior to this study.
13. Subject is taking >10 mg prednisone (or equivalent dose of a similar steroid) daily.
14. Subject requires high level chronic immunomodulatory therapy to treat a moderate to severe chronic inflammatory autoimmune disorder.
15. Subject is on an antiplatelet (such as Plavix) or anticoagulant therapy (such as heparin or Coumadin) which cannot be stopped prior to procedure.
16. Subject has a known sensitivity or allergy to Nickel
17. Subject has a known sensitivity to drugs required to perform bronchoscopy.
18. Subject has any other disease, condition(s) or habit(s) that would interfere with completion of study and follow up assessments, would increase risks of bronchoscopy or assessments, or in the judgment of the investigator would potentially interfere.
19. Alfa-1 AT deficiency
20. Medical history of asthma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-03; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in physical activity at 3 months. | Baseline vs 3 months follow up
  *Change in physical activity measured by an accelerometer, 3 months following treatment.

SECONDARY OUTCOMES:
Change from baseline in patient reported outcomes of the treatment at 3 months follow up. | Baseline vs 3 months follow up
  *Change in patient reported outcomes measured by the PSK (Patient Specifieke Klachten)-questionnaire, 3 months following treatment.
Change from baseline in dynamic lung hyperinflation at 3 months follow up. | Baseline vs 3 months follow up
  * Change in dynamic hyperinflation measured by a metronome-paced tachypnea test, 3 months following treatment.
  * Change in dynamic hyperinflation measured by a maximum incremental cycle ergometer test, 3 months following treatment.
  * Change in inspiratory capacity (IC) measurement before and after the 6-minute walk distance test, 3 months following treatment.
Change from baseline in static lung volumes at 3 months follow up. | Baseline vs 3 months follow up
  * Change in lung volumes measured by bodyplethysmography, 3 months following treatment.
  * Change in lung volumes measured using HRCT analysis, 3 months following treatment.
Change from baseline in lung compliance at 3 months follow up. | Baseline vs 3 months follow up
  *Change in lung compliance measured by a balloon catheter system, 3 months following treatment.
Change from baseline in diaphragm function at 3 months follow up. | Baseline vs 3 months follow up.
  *Change in diaphragm function measured by inspiratory and expiratory muscle strength (PI-max & PE-max), 3 months following treatment.
Change from baseline in lung perfusion at 3 months follow up. | Baseline vs 3 months follow up.
  *Change in quantified lung perfusion assessment measured by a perfusion scan using 99mTc albumin, 3 months following treatment.
Change from baseline in small airways function at 3 months follow up. | Baseline vs 3 months follow up
  * Change in air trapping scores of in-and expiratory HRCT scan analysis, 3 months following treatment.
  * Change in multiple breath nitrogen N2-washout (up to 1/20) measurement, 3 months following treatment.
Change from baseline in systemic inflammation at 3 months follow up. | Baseline vs 3 months follow up
  *Change in systemic inflammation markers measured in blood (hs-CRP, IL-6, IL-8, TNFα, fibrinogen), 3 months following treatment.

OTHER OUTCOMES:
Identification of Responders | Baseline vs 3 months follow up
  *Association between baseline characteristics and outcome variables 3 months after the second treatment to try to identify responders and non responders.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk-Jan Slebos, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- University Medical Center Groningen, Groningen, Netherlands
- Royal Brompton Hospital & Imperial College, London, United Kingdom